CLINICAL TRIAL: NCT07376525
Title: Comparison of the Effects of Percutaneous Dilatational Tracheostomy Performed With Fiberoptic Bronchoscopy and Ultrasound Guidance on Ventilation
Brief Title: Comparison of Ventilatory Effects of Ultrasound-Guided Versus Bronchoscopy-Guided Percutaneous Dilatational Tracheostomy
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Rabia Sarı Küçük, Intensive Care Specialist, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Other Study IDs: CT-ERHO-AR-BA-02
Record Dates: First submitted 2026-01-22; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Respiratory Failure; Mechanical Ventilation; Tracheostomy
Keywords: Percutaneous Dilatational Tracheostomy; Fiberoptic Bronchoscopy; Ultrasonography; Mechanical Ventilation; Intensive Care Unit; Arterial Blood Gas; Ventilation Parameters
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fiberoptic Bronchoscopy-Guided Percutaneous Dilatational Tracheostomy: Adult ICU patients who underwent percutaneous dilatational tracheostomy guided by fiberoptic bronchoscopy as part of routine clinical practice.
  Interventions: Procedure: Percutaneous Dilatational Tracheostomy Guidance Method
- Ultrasonography-Guided Percutaneous Dilatational Tracheostomy: Adult ICU patients who underwent percutaneous dilatational tracheostomy guided by ultrasonography as part of routine clinical practice.
  Interventions: Procedure: Percutaneous Dilatational Tracheostomy Guidance Method

INTERVENTIONS:
Procedure: Percutaneous Dilatational Tracheostomy Guidance Method — Percutaneous dilatational tracheostomy performed under either fiberoptic bronchoscopy or ultrasonography guidance according to routine clinical practice. No interventions were assigned by study protocol.

SUMMARY:
Percutaneous dilatational tracheostomy (PDT) is a commonly performed procedure in intensive care units for patients requiring prolonged mechanical ventilation. Fiberoptic bronchoscopy (FOB) and ultrasonography (USG) are frequently used to guide PDT in order to improve procedural safety. However, the effects of these guidance techniques on ventilation parameters during the procedure remain unclear.

This retrospective observational study aims to compare the effects of FOB-guided and USG-guided percutaneous dilatational tracheostomy on ventilation parameters in mechanically ventilated adult intensive care unit patients. Changes in arterial blood gas parameters and ventilator settings during and after the procedure will be evaluated.

The findings of this study may help clinicians better understand the physiological effects of different PDT guidance techniques and support informed decision-making in clinical practice.

DETAILED DESCRIPTION:
Percutaneous dilatational tracheostomy (PDT) is widely used in intensive care units (ICUs) as an alternative to surgical tracheostomy in patients requiring prolonged mechanical ventilation. Various guidance methods have been introduced to increase procedural safety and accuracy, including fiberoptic bronchoscopy (FOB) and ultrasonography (USG). While both techniques are commonly used, their effects on ventilation and gas exchange during the procedure are still debated.

Fiberoptic bronchoscopy allows direct visualization of the tracheal lumen and needle placement but may partially obstruct the airway, potentially leading to increased airway pressures, hypercapnia, and impaired ventilation. Ultrasonography, on the other hand, enables real-time visualization of neck anatomy without entering the airway and may therefore have different effects on ventilation parameters.

This retrospective observational study includes adult ICU patients who underwent percutaneous dilatational tracheostomy between May 5, 2023, and September 1, 2025. Patients were grouped according to the guidance technique used during the procedure: FOB-guided PDT or USG-guided PDT. All procedures were performed under standard ICU conditions by experienced clinicians.

Demographic data, clinical characteristics, ventilator settings, and arterial blood gas parameters were collected from patient records. Primary outcomes included changes in arterial blood gas values (pH, PaCO₂, PaO₂) and ventilatory parameters before, during, and after the procedure. Secondary outcomes included procedure duration and procedure-related complications.

The study aims to compare the effects of FOB-guided and USG-guided PDT on ventilation and gas exchange, providing insight into the physiological consequences of each technique. As a retrospective observational study, no additional interventions were performed beyond standard clinical practice.

The results of this study may contribute to optimizing guidance method selection during percutaneous dilatational tracheostomy and improving patient safety in the intensive care setting.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (≥18 years of age) Patients admitted to the intensive care unit Patients receiving invasive mechanical ventilation Patients who underwent percutaneous dilatational tracheostomy under fiberoptic bronchoscopy or ultrasonography guidance Availability of complete clinical and arterial blood gas data

Exclusion Criteria:

Age <18 years Patients with incomplete medical records or missing arterial blood gas data Patients who underwent surgical (open) tracheostomy Patients with pre-existing tracheal pathology affecting ventilation parameters

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult intensive care unit patients who required prolonged invasive mechanical ventilation and underwent percutaneous dilatational tracheostomy guided by either fiberoptic bronchoscopy or ultrasonography as part of routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2025-09-15 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Change in Ventilation and Arterial Blood Gas Parameters During Percutaneous Dilatational Tracheostomy | Immediately before the procedure, during the procedure, and immediately after the procedure
  Changes in arterial blood gas parameters (pH, PaCO₂, PaO₂) and ventilatory parameters measured before, during, and after percutaneous dilatational tracheostomy, comparing fiberoptic bronchoscopy-guided and ultrasonography-guided procedures.

SECONDARY OUTCOMES:
Procedure Duration | During the procedure
  Total duration of the percutaneous dilatational tracheostomy procedure, measured from skin incision to successful tracheostomy tube placement.
Procedure-Related Complications | During the procedure and the immediate post-procedural period
  Incidence of procedure-related complications, including hypoxia, hypercapnia, bleeding, hypotension, pneumothorax, and other clinically relevant adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization, Istanbul, Sisli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No